CLINICAL TRIAL: NCT05554835
Title: Global Mitochondrial Registry to Define Natural History and Outcome Measures to Achieve Definite Trial Readiness for Mitochondrial Disorders
Brief Title: Global Registry and Natural History Study for Mitochondrial Disorders
Acronym: GENOMIT
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: European Commission (Other); German Federal Ministry of Education and Research (Other Government); University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Thomas Klopstock, Prof. Dr. Thomas Klopstock, LMU Klinikum
Other Study IDs: mitoGLOBAL
Record Dates: First submitted 2022-08-11; First posted 2022-09-26 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Mitochondrial Diseases; Kearns-Sayre Syndrome; MIDD; SANDO; SCAE; NARP Syndrome; MELAS Syndrome; MERRF Syndrome; Coenzyme Q10 Deficiency; LHON; MNGIE; MIRAS; Barth Syndrome; MDS; Mitochondrial Myopathies; Leigh Syndrome; Pearson Syndrome; CPEO
Keywords: Patient Registry
MeSH Terms: conditions — Mitochondrial Diseases; Kearns-Sayre Syndrome; Ataxia Neuropathy Spectrum; Neuropathy ataxia and retinitis pigmentosa; MELAS Syndrome; MERRF Syndrome; Coenzyme Q10 Deficiency; Barth Syndrome; Mitochondrial Myopathies; Leigh Disease; VLCAD deficiency; Ophthalmoplegia, Chronic Progressive External

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mitochondrial patients: Patients with a suspected or confirmed mitochondrial disease.

SUMMARY:
The main goal of the project is provision of a global registry for mitochondrial disorders to harmonize previous national registries, enable world-wide participation and facilitate natural history studies, definition of outcome measures and conduction of clinical trials.

DETAILED DESCRIPTION:
The global mitochondrial registry and natural history study is part of the EU-financed GENOMIT project, co-ordinated by Dr. Holger Prokisch, Technische Universität München (TUM).It aims at advancing the understanding of the natural history of mitochondrial disease to inform the design and facilitate the conduction of clinical trials. It also serves as a catalyst for translating basic research results into clinical practice.

The global mitochondrial registry and natural history study provides for all contingencies of national ethics and data protection rules including data access management.

Currently participating networks are:

* German network for mitochondrial diseases - mitoNET, Germany/Austria
* Italian Registry of Mitochondrial Patients - Mitocon, Italy

The inclusion of other networks and countries is possible and explicitly welcome. A major advantage of the global registry is that countries can join in, saving a lot of time, effort and funding.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed mitochondrial disease
* willingness to participate

Exclusion Criteria:

* unwillingness to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2009-02-01 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Newcastle Mitochondrial Disease Scale for Adults (NMDAS), Sections I-III | The individual participants are followed with annual assessments over a long time period (up to 30 years) or until discontinuation or death.
  Newcastle Mitochondrial Disease Scale for Adults (NMDAS) is a clinical rating scale designed for mitochondrial disease. The rating scale explores several domains: current function, system specific involvement and current clinical assessment. The individual scores are summed to provide a total score that ranges from 0 to 145; higher scores indicate more severely affection.
Newcastle Pediatric Mitochondrial Disease Scale for Children (NPMDS) | The individual participants are followed with annual assessments until they reach the next age group version (up to 18 years) or until discontinuation or death.
  NPMDS is a clinical rating scale designed for mitochondrial disease in children.
  There are three versions of the NPMDS, each for a specific age range (0-24 months, 2-11 years, and 12-18 years). The rating scale explores several domains: current function (Section I), system specific involvement (Section II), current clinical assessment (Section III) and quality of life (QoL) assessments (Section IV). The individual scores in Section I-III are summed to provide a total score that ranges from 0 to 70 (version 0-24month) and 0-82 (versions 2-18 years); higher scores indicate more severely affection. Section IV (QoL) is scored separately and provide a total score that ranges from 0 to 25 with higher scores indicating better quality of life.
Scale for the assessment and rating of ataxia (SARA) in adults | The individual participants are followed with annual assessments over a long time period (up to 30 years) or until discontinuation or death.
  The Scale for the Assessment and Rating of Ataxia (SARA) is a clinical scale used to assess cerebellar ataxia in adults. The scale includes 8 items, related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test. The individual scores are summed to provide a total score that ranges from 0 to 40, higher scores indicate more severe ataxia.
Disease progression | The individual participants are followed with annual assessments over a long time period (up to 30 years) or until discontinuation or death.
  Disease progression as assessed by clinical examination and captured as HPO (Human Phenotype Ontology) Terms at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klopstock, Prof. Dr., Principal Investigator — LMU Klinikum, Munich; Michelangelo Mancuso, Prof. Dr., Principal Investigator — Università di Pisa
Locations (18):
- Austria (2):
  - Medical University Innsbruck, Department of Pediatrics, Innsbruck
  - Salzburger Landeskliniken, SALK, Paracelsus Medizinische Privatuniversität, Salzburg
- Germany (15):
  - Department of neurology, Klinikum rechts der Isar, Technical University Munich, Munich, Bavaria
  - Charité Virchow Klinikum, Klinik für Pädiatrie m. S. Neurologie, Berlin
  - Universität Bonn, Klinik und Poliklinik für Neurologie, Bonn
  - Universitätsklinikum Köln, Klinik und Poliklinik für Kinder- und Jugendmedizin, Cologne
  - Universitätsklinikum Düsseldorf, Klinik für allgemeine Pädiatrie, Neonatologie und Kinderkardiologie, Düsseldorf
  - Universitätsklinikum Frankfurt, Klinik für Kinder- und Jugendmedizin, Schwerpunkt Neurologie, Neurometabolik und Prävention, Frankfurt am Main
  - University Medical Center Freiburg, Center for children and youth medicine, Freiburg im Breisgau
  - Martin-Luther-Universität Halle-Wittenberg, Neurologische Klinik und Poliklinik, Halle
  - Universitätsklinikum Hamburg Eppendorf Institut für Humangenetik, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Klinik für Kinder-und Jugendmedizin, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Klinik für Neurologie, Hamburg
  - Universitätsklinikum Heidelberg, Zentrum für Kinder- und Jugendmedizin, Sektion für Neuropädiatrie und Stoffwechselmedizin, Heidelberg
  - LMU Klinikum, Friedrich-Baur-Institut an der Neurologischen Klinik und Poliklinik, München
  - Klinikum am Steinenberg, Kreiskliniken Reutlingen, Klinik für Kinder-und Jugendmedizin, Perinatal- u. Stoffwechselzentrum, Reutlingen
  - Universitätsklinikum Tübingen, Neurologische Klinik und Hertie Institut für Klinische Hirnforschung, Tübingen
- Department of Clinical and Experimental Medicine, Neurological Institute, University of Pisa & AOUP, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
Any data or results from the project can be shared upon written request with researchers. Data sharing requires approval by the respective scientific committee and their institutional review board.
Supporting Information: ICF
Time Frame: Time frame for data usage needs to be specified in the proposal for data sharing.
Access Criteria: Approved written proposal including the description of the research plan and data usage purpose.
URL: https://www.mitonet.org/netzwerk/patientenregister_biobank/beantragung-von-daten-proben/

REFERENCES:
- [Background] Stenton SL, Sheremet NL, Catarino CB, Andreeva NA, Assouline Z, Barboni P, Barel O, Berutti R, Bychkov I, Caporali L, Capristo M, Carbonelli M, Cascavilla ML, Charbel Issa P, Freisinger P, Gerber S, Ghezzi D, Graf E, Heidler J, Hempel M, Heon E, Itkis YS, Javasky E, Kaplan J, Kopajtich R, Kornblum C, Kovacs-Nagy R, Krylova TD, Kunz WS, La Morgia C, Lamperti C, Ludwig C, Malacarne PF, Maresca A, Mayr JA, Meisterknecht J, Nevinitsyna TA, Palombo F, Pode-Shakked B, Shmelkova MS, Strom TM, Tagliavini F, Tzadok M, van der Ven AT, Vignal-Clermont C, Wagner M, Zakharova EY, Zhorzholadze NV, Rozet JM, Carelli V, Tsygankova PG, Klopstock T, Wittig I, Prokisch H. Impaired complex I repair causes recessive Leber's hereditary optic neuropathy. J Clin Invest. 2021 Mar 15;131(6):e138267. doi: 10.1172/JCI138267. PMID 33465056
- [Background] Stendel C, Neuhofer C, Floride E, Yuqing S, Ganetzky RD, Park J, Freisinger P, Kornblum C, Kleinle S, Schols L, Distelmaier F, Stettner GM, Buchner B, Falk MJ, Mayr JA, Synofzik M, Abicht A, Haack TB, Prokisch H, Wortmann SB, Murayama K, Fang F, Klopstock T; ATP6 Study Group. Delineating MT-ATP6-associated disease: From isolated neuropathy to early onset neurodegeneration. Neurol Genet. 2020 Jan 13;6(1):e393. doi: 10.1212/NXG.0000000000000393. eCollection 2020 Feb. PMID 32042921
- [Background] Ng YS, Bindoff LA, Gorman GS, Klopstock T, Kornblum C, Mancuso M, McFarland R, Sue CM, Suomalainen A, Taylor RW, Thorburn DR, Turnbull DM. Mitochondrial disease in adults: recent advances and future promise. Lancet Neurol. 2021 Jul;20(7):573-584. doi: 10.1016/S1474-4422(21)00098-3. PMID 34146515
- [Background] Ng YS, Bindoff LA, Gorman GS, Horvath R, Klopstock T, Mancuso M, Martikainen MH, Mcfarland R, Nesbitt V, Pitceathly RDS, Schaefer AM, Turnbull DM. Consensus-based statements for the management of mitochondrial stroke-like episodes. Wellcome Open Res. 2019 Dec 13;4:201. doi: 10.12688/wellcomeopenres.15599.1. eCollection 2019. PMID 32090171
- [Background] Mancuso M, McFarland R, Klopstock T, Hirano M; consortium on Trial Readiness in Mitochondrial Myopathies. International Workshop:: Outcome measures and clinical trial readiness in primary mitochondrial myopathies in children and adults. Consensus recommendations. 16-18 November 2016, Rome, Italy. Neuromuscul Disord. 2017 Dec;27(12):1126-1137. doi: 10.1016/j.nmd.2017.08.006. Epub 2017 Sep 8. No abstract available. PMID 29074296
- See also: Project website — https://genomit.eu/work-packages/global-registry-and-trial-readiness/index.html
- See also: mitoNET website — https://www.mitonet.org/netzwerk/patientenregister_biobank/
- See also: Mitocon website — https://www.mitocon.it/